CLINICAL TRIAL: NCT01016964
Title: A Randomized, Double-Blind Clinical Trial to Evaluate the Safety and Efficacy of the HairMax LaserComb 2009, 12 Beam Model For The Treatment of Androgenetic Alopecia in Females
Brief Title: Treatment of Androgenetic Alopecia in Females, 12 Beam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lexington International, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12 2009-F-02; NCT01042756 (obsolete NCT alias)
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-08

CONDITIONS: Androgenetic Alopecia; Hair Loss; Female Pattern Baldness
Keywords: Androgenetic Alopecia; Hair Loss; Female Pattern Baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham Device (Sham Comparator): Sham device
  Interventions: Device: Sham Device
- LLT Device 2009 12 Beams (Active Comparator): HairMax LaserComb 2009 model 12 beam
  Interventions: Device: HairMax LaserComb 2009 model 12 beam

INTERVENTIONS:
Device: HairMax LaserComb 2009 model 12 beam — HairMax LaserComb
  Arms: LLT Device 2009 12 Beams
Device: Sham Device — Sham Device
  Arms: Sham Device

SUMMARY:
The purpose of this study is to evaluate the efficacy of the HairMax LaserComb 2009 12 beam model for androgenetic alopecia in females when treatment is applied as directed.

DETAILED DESCRIPTION:
This is a randomized double-blind, sham controlled clinical study, evaluating changes in terminal hair count in the evaluation zone having evidence of androgenetic alopecia (miniaturized hair).

The trial with 63 female subjects, who have been diagnosed with androgenetic alopecia, who are between 25 and 60 years of age, have Fitzpatrick Skin Types I-IV, with classifications of Ludwig I-4, II-1, II-2, or frontal, have active hair loss within the last 12 months.

Subjects will use the device on three non-concurring days a week as directed per device for 26 weeks duration.

Initial efficacy endpoint for each subject will be assessed at visit 4 (week 16).

Safety analysis will be assessed based on the reports of adverse events during study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of androgenetic alopecia
* Fitzpatrick Skin types I-IV
* Ludwig I-4, II-1, II-2, or frontal
* Active hair loss within last 12 months

Exclusion Criteria:

* Photosensitivity to laser light
* Malignancy in the target area
* Pregnancy
* Lactating females

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, M.D., Principal Investigator — University of Minnesota; Wilma Bergfeld, M.D., Principal Investigator — The Cleveland Clinic; Lawrence Schachner, M.D., Principal Investigator — University of Miami
Locations (3):
- United States (3):
  - University of Miami Miller School of Medicine - Dermatology, Miami, Florida
  - University of Minnesota, Department of Dermatology, Minneapolis, Minnesota
  - Cleveland Clinic Foundation - Department of Dermatology, Cleveland, Ohio

REFERENCES:
- [Background] Leavitt M, Charles G, Heyman E, Michaels D. HairMax LaserComb laser phototherapy device in the treatment of male androgenetic alopecia: A randomized, double-blind, sham device-controlled, multicentre trial. Clin Drug Investig. 2009;29(5):283-92. doi: 10.2165/00044011-200929050-00001. PMID 19366270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This double-blind, device controlled 26 week study was recruited at 3 clinical study sites. The recruitment period was from February 1, 2010 to September 28, 2010
Pre-assignment Details: Key exclusion criteria was pregnancy, malignancy in target area, an no hair transplants, scalp reductions, or hair weaves. Active hair loss less than 12 months.
Period: Overall Study
Arm/Group | Sham Device | LLT Device 2009 12 Beams
Started | 21 | 42
Completed | 18 | 39
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Device | LLT Device 2009 12 Beams | Total
Number analyzed (Participants) | 21 | 42 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 42 | 63
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 42 | 63
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Hair Count at 16 and 26 Weeks Over Baseline
Description: The primary analysis of effectiveness was an analysis of covariance, which separately modeled terminal hair count at Week 16 and Week 26 as a function of treatment group (HairMax LaserComb 2009 9 Beam vs.control), study center, age (as a continuous variable), and Fitzpatrick Skin Type classification (as a categorical variable with four levels). The active group was compared to the control device using least squares means with a two-sided test at the 5% level of significance.
Time Frame: Baseline, 16 weeks, 26 weeks
Measure: Mean (Standard Deviation); unit: hairs per cm^2
Groups:
- Sham Device: This control device emits white light
- LLT Device 2009 12 Beams: This is the active LLLT device
Arm/Group | Sham Device | LLT Device 2009 12 Beams
Number analyzed (Participants) | 18 | 39
hairs per cm^2
  Change at 16 weeks | -0.8 (7.87) | 12.5 (11.35)
  Change at 26 weeks | 3.0 (9.33) | 20.6 (11.55)

ADVERSE EVENTS:
Arm/Group | Sham Device | LLT Device 2009 12 Beams
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/39
Other Adverse Events (participants affected / at risk) | 0/18 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No